CLINICAL TRIAL: NCT07271459
Title: Effect of Propofol and Dexmedetomidine-Based Total Intravenous Anesthesia Versus Sevoflurane-Based Inhalational Anesthesia on the Level of Inflammatory Markers in Patients Undergoing Inguinal Hernia Repair.
Brief Title: Effect of Total Intravenous Anesthesia vs Inhalational Anesthesia on the Level of Inflammatory Markers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MD256/2025
Record Dates: First submitted 2025-11-13; First posted 2025-12-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: Anesthesia
Keywords: TIVA; Inhalational Anesthesia; Inflammatory Markers
MeSH Terms: interventions — Propofol; Dexmedetomidine; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Collector of blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIVA group (group A) in which both propofol and dexmedetomidine will be used together (Active Comparator): Group A (TIVA group): will receive 1 μg/kg IV dexmedetomidine over 10 min, 1 μg/kg IV fentanyl, 2 mg/kg IV propofol, and 0.5 mg/kg IV atracurium. Maintenance of anesthesia will be achieved by 0.5 μg/kg/h dexmedetomidine IV infusion and 6-12 mg/kg/h propofol IV infusion titrated according to bispectral index value (BIS) with target BIS 40-60.
  Interventions: Diagnostic Test: Venous blood sampling preoperatively; Diagnostic Test: Venous blood sampling at 6 hours postoperative; Diagnostic Test: Venous blood sampling at 24 hours postoperative; Drug: Propofol; Drug: Dexmedetomidine
- Sevoflurane group (group B) (Active Comparator): Group B (Sevoflurane group): will receive 1 μg/kg IV fentanyl, 8% sevoflurane via face mask and 0.5 mg/kg IV atracurium. Maintenance of anesthesia will be achieved with 2%-4% sevoflurane titrated according to BIS with target BIS 40-60
  Interventions: Diagnostic Test: Venous blood sampling preoperatively; Diagnostic Test: Venous blood sampling at 6 hours postoperative; Diagnostic Test: Venous blood sampling at 24 hours postoperative; Drug: Sevoflurane

INTERVENTIONS:
Diagnostic Test: Venous blood sampling preoperatively — 5 mL of venous blood will be aseptically withdrawn into a sterile plain tube. Serum interleukin-6 (IL-6) levels will be measured using the enzyme-linked immunosorbent assay (ELISA) method.
  Ferritin and C-reactive protein (CRP) concentrations will be analyzed using a COBAS automated analyzer.
  Additionally, a 2 mL blood sample will be collected in an EDTA tube for complete blood count (CBC) analysis, which will be performed using the Sysmex Coulter hematology analyzer
Diagnostic Test: Venous blood sampling at 6 hours postoperative — 5 mL of venous blood will be aseptically withdrawn into a sterile plain tube. Serum interleukin-6 (IL-6) levels will be measured using the enzyme-linked immunosorbent assay (ELISA) method.
  Ferritin and C-reactive protein (CRP) concentrations will be analyzed using a COBAS automated analyzer.
  Additionally, a 2 mL blood sample will be collected in an EDTA tube for complete blood count (CBC) analysis, which will be performed using the Sysmex Coulter hematology analyzer
Diagnostic Test: Venous blood sampling at 24 hours postoperative — 5 mL of venous blood will be aseptically withdrawn into a sterile plain tube. Serum interleukin-6 (IL-6) levels will be measured using the enzyme-linked immunosorbent assay (ELISA) method.
  Ferritin and C-reactive protein (CRP) concentrations will be analyzed using a COBAS automated analyzer.
  Additionally, a 2 mL blood sample will be collected in an EDTA tube for complete blood count (CBC) analysis, which will be performed using the Sysmex Coulter hematology analyzer
Drug: Propofol — Group A (TIVA group): will receive 1 μg/kg IV dexmedetomidine over 10 min, 1 μg/kg IV fentanyl, 2 mg/kg IV propofol, and 0.5 mg/kg IV atracurium. Maintenance of anesthesia will be achieved by 0.5 μg/kg/h dexmedetomidine IV infusion and 6-12 mg/kg/h propofol IV infusion titrated according to bispectral index value (BIS) with target BIS 40-60.
  Arms: TIVA group (group A) in which both propofol and dexmedetomidine will be used together
Drug: Dexmedetomidine — Group A (TIVA group): will receive 1 μg/kg IV dexmedetomidine over 10 min, 1 μg/kg IV fentanyl, 2 mg/kg IV propofol, and 0.5 mg/kg IV atracurium. Maintenance of anesthesia will be achieved by 0.5 μg/kg/h dexmedetomidine IV infusion and 6-12 mg/kg/h propofol IV infusion titrated according to bispectral index value (BIS) with target BIS 40-60.
  Arms: TIVA group (group A) in which both propofol and dexmedetomidine will be used together
Drug: Sevoflurane — Group B (Sevoflurane group): will receive 1 μg/kg IV fentanyl, 8% sevoflurane via face mask and 0.5 mg/kg IV atracurium. Maintenance of anesthesia will be achieved with 2%-4% sevoflurane titrated according to BIS with target BIS 40-60
  Arms: Sevoflurane group (group B)

SUMMARY:
This study aims to compare the effects of total intravenous anesthesia (TIVA) vs inhalational anesthesia on postoperative levels of inflammatory markers, length of hospital stay, and the incidence of postoperative nausea and vomiting in patients undergoing inguinal hernia repair.

Number participants:

Participants will be divided into 2 groups with sample size of at least 20 patients per group.

Plan of the work:

All patients will receive general anesthesia according to Ain Shams hospital protocol which follows the standards of the American Society of Anesthesiologists. Group A will be TIVA group and Group B will be Sevoflurane group.

Sample Collection and Laboratory Analysis:

Venous blood samples will be collected from each patient at three time points:

preoperative (baseline, sample 0), 6 hours postoperative (sample 1), and 24 hours postoperative (sample 2).

DETAILED DESCRIPTION:
Aim of study: Several studies showed that the anesthetic technique can affect several postoperative outcomes including the level of inflammatory markers such as Interleukins (ILs), C-reactive protein (CRP), ferritin, and neutrophil-to-lymphocyte ratio (NLR). This study aims to compare the postoperative levels and trends of change of inflammatory markers, namely IL-6, CRP, ferritin, and NLR in patients undergoing inguinal hernia repair using propofol and dexmedetomidine-based total intravenous anesthesia (TIVA) vs sevoflurane-based inhalational anesthesia (IA).

Type of Study: Prospective, randomized, double-blind, comparative clinical study.

Study Setting: Ain Shams University hospitals, Cairo, Egypt. Study Period: 6-12 months. Study Population: Adult patients scheduled for elective inguinal hernia repair. Sampling Method: Random sampling Sample Size: Using the PASS 15 program from sample size calculation, reviewing results from the previous study (Yediyıldız et al., 2025) showed that postoperative IL-6 levels were significantly lower in the TIVA group than in the sevoflurane group 20,1±23,5 versus 54,8±45,4, based on these findings a sample size of at least 20 patients per group achieve 80% power to reject the null hypothesis of equal means when the population mean difference is μ1-μ2 = 54.8- 4 20.1 = 34.7 with standard deviations of 45.0 for group 1 and 23.5 for group 2, and with a significance level (alpha) of 0.050 using a two-sided two-sample unequal-variance t-test. Ethical Considerations: The study protocol received ethical approval from the Research Ethical Committee, Faculty of Medicine Ain Shams University. Written informed consent will be signed by all participants before starting study.

Randomization and blinding: Group allocation will be contained in sequentially numbered, sealed opaque envelopes, which will be opened by the primary investigator. The collector of blood samples and the data analyzer will be blinded about the study group.

Study Procedures:

All patients will be assessed preoperatively by careful history taking and airway examination. Complete blood count (CBC), coagulation profile, liver and kidney function tests for all patients and electrocardiogram (ECG) for patients older than 40 years of age will be reviewed from patients medical records. All patients will be admitted after completing fasting hours for both solid food and clear fluids. Upon arrival to the operating room (OR), IV access of the size 20 gauge (G) will be inserted. All patients will be monitored with a five-lead ECG, non-invasive blood pressure (NIBP) measurement and finger pulse oximetry. Baseline vital data (MAP, HR, and oxygen saturation (SO2)) will be recorded. HR and SO2 will be monitored continuously and BP will be measured every 5 minutes (min) till the end of the surgery.

All patients will be premedicated with 0.03 mg/kg IV midazolam. Preoxygenation will be performed using 100% oxygen at a fresh gas flow (FGF) of 10 L/min via face mask for 3 minutes, followed by induction of general anesthesia.

Detailed anesthetic technique followed with both groups (TIVA group and Sevoflurane group) will be mentioned in arms and interventions section.

After induction, intubation will be done for all patients using suitable size endotracheal tube (ETT). Both groups will be mechanically ventilated using volume control mode with tidal volume 7-10 ml/kg/min, positive end-expiratory pressure (PEEP) 5 cmH2O and oxygen-air mixture with fraction of inspired oxygen (FiO2) 50% and FGF of 3 L/min, and respiratory rate adjusted with target end-tidal carbon dioxide (ET CO2) 30-40 mmHg. 0.1 mg/kg IV atracurium will be given as needed to maintain muscle relaxation. 0.5 mcg/kg fentanyl will be given if HR or MAP increase ≥20% from their basal value. HR and MAP ≤20% of the basal value will be treated with needed doses of atropine and ephedrine, respectively. All patients will be extubated in the operating room and transferred to postanesthesia care unit (PACU).

Sample Collection and Laboratory Analysis:

Venous blood samples for IL-6, CRP, ferritin, and CBC will be collected from each patient at three time points: preoperative (baseline, sample 0), 6 hours postoperative (sample 1), and 24 hours postoperative (sample 2). All laboratory analysis will be conducted at the main laboratories of Ain Shams University Hospital.

❖ The main researcher of the study will be the principal investigator responsible for the preparation and conduct of the study under supervision of the director and co-directors. Each member of the team will ensure that the study is conducted according to the protocol approved in their meetings that will be arranged on regular basis. Results of the study and any complications that might occur during the study will be recorded and reported by the principal investigator and revised by the director and co-directors. Statistical Analysis The collected data will be revised, coded and introduced to a PC using statistical package for social science (SPSS 23).

Data will be presented as mean and standard deviation (+/-SD) for quantitative parametric data, median and range for quantitative non-parametric data and as numbers and percentage for qualitative data. Suitable analysis will be done according to the type of data obtained. P< 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients between 18 and 50 years of age undergoing elective inguinal hernia repair.
2. American Society of Anesthesiologists physical status classification (ASA) I and II.

Exclusion Criteria:

1. Patient's refusal.
2. ASA > II
3. Complicated hernia.
4. Previous hernia repair with mesh.
5. History of allergy to any of the study drugs.
6. History of any heart disease affecting cardiac function or rhythm or receiving medications that decrease the heart rate (HR).
7. Baseline HR≤60 beat/min.
8. Baseline mean arterial pressure (MAP)≤70 mmHg.
9. Psychiatric illness.
10. Patients with chronic kidney or liver disease. (Creatinine clearance<50 mL/min or serum albumin level<2g/dL.)
11. Patients with immunological disorders or receiving immunosuppressive treatment or anti-inflammatory drugs.
12. Patients with neoplasms, chronic inflammatory states, or active infections.
13. Patients with any type of anemia or those who received iron therapy or blood transfusion within 4 weeks.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
IL-6 level 24 hours postoperatively compared to baseline value | 24 hours
  Venous blood samples will be withdrawn aseptically at 3 time points (preoperative, 6 hours postoperative, and 24 hours postoperative)

SECONDARY OUTCOMES:
Trend of change of IL-6 level within the postoperative 24 hours. | 24 hours
  Venous blood samples will be withdrawn aseptically at 3 time points for the level of inflammatory markers and patients' medical records will be reviewed for the rest of the outcomes
Trends of change and levels of CRP, NLR, and ferritin 24 hours postoperatively. | 24 hours
  Venous blood samples will be withdrawn aseptically at 3 time points for the level of inflammatory markers.
Time to discharge. | 24 hours
  patients' medical records will be reviewed.
Incidence of PONV. | 24 hours
  patients' medical records will be reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Doha A Elgamal, MBBCh, MSc, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the study results will be made available upon reasonable request from qualified researchers.
Supporting Information: Study Protocol
Time Frame: Within 6-12 months and for up to 5 years
Access Criteria: Access will be granted to researchers who submit a methodologically sound proposal to the principal investigator. Requests should be directed to dohaatef@med.asu.edu.eg

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT07271459/Prot_SAP_000.pdf